Study's Official Title: Effectiveness of a Mobile Texting Intervention for People with Serious Mental

Illness

NCT Number: NCT03062267

Date of Document: 10/9/2020

<u>Document Title:</u> Study Protocol with Statistical Analysis Plan

## **Study Protocol**

We conducted an assessor-blind, two-arm, randomized controlled trial in partnership with assertive community treatment (ACT) teams providing services to individuals with serious mental illness in the Midwest and Pacific Northwest regions of the United States. The research was monitored by an independent safety monitoring board at the University of Washington's School of Medicine. Participants provided informed consent. All participants were receiving ACT services and were randomly assigned to one of two treatment arms: mobile interventionist (ACT augmented with mobile phone texting) or treatment as usual (standard ACT). Interventions were deployed for 3 months. We conducted assessments at baseline (0 months), posttrial (3 months), and follow-up (6 months). Participants were compensated for completing assessments (\$30 per assessment, plus reimbursement for travel).

## Statistical Analysis Plan

Primary outcomes will be assessed by change in means and standard deviations of measures used. Secondary outcomes will be assessed by change in means and standard deviations of measures used. The other pre-specified outcome measure of Satisfaction with Treatment at 3 months following intervention period will be assessed by evaluating means and standard deviations, and comparing the intervention group to the control group.